CLINICAL TRIAL: NCT03907709
Title: Effects of an In-Home Treatment Program for First Responders With Substance Use Disorder: A Retrospective Analysis
Brief Title: Effects of In-Home Addiction Treatment for First Responders
Status: Suspended | Type: Observational
Why Stopped: Resource allocation
Sponsor: In-Home Addiction Treatment Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IHATI-2019-1
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First Responders in In-Home Addiction Treatment Program: - First responders (individual who does or has worked as a police officer, fire fighter, corrections officer, military police, emergency medical technician, paramedic, parole or probation officer)
  Interventions: Behavioral: In-Home Addiction Treatment Program

INTERVENTIONS:
Behavioral: In-Home Addiction Treatment Program — * Treatment was delivered per treatment protocol
  * Primary IHAT Care Team consisted of a licensed Care Coordinator (LPN, RN, MSW, LPC, or LMFT) and two Recovery Advisors
  * Urine drug screens administered randomly
  * Appointments were scheduled per protocol for 52 weeks
  * Within first two weeks of care, all clients are provided an evaluation by a psychiatrist to ensure fitness for program

SUMMARY:
Retrospective analysis to evaluate impact of an in-home addiction treatment program on first responders with substance use disorder.

DETAILED DESCRIPTION:
The purpose of this retrospective study is to evaluate the effects of in-home addiction treatment on first responders with substance use disorder. Treatment engagement, hospitalizations, detox and residential addiction treatment admissions, and lethal overdoses will be measured. Although not the primary focus, recidivism and relapse will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Client is or has been a first responder
* Client enrolled in Aware Recovery Care after April 2017
* Client discharged from Aware Recovery Care before March 2019
* Client has primary substance use disorder diagnosis

Exclusion Criteria:

* Client has never been first responder
* Client moved out of service area or lost insurance during care

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 15 individuals with substance use disorder who are or have served as a first responder (police officer, fire fighter, corrections officer, military police, emergency medical technician, paramedic, parole or probation officer) and were enrolled in Aware Recovery Care's In-Home Addiction Treatment program between April 2017 and March 2019.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-05-28 (Estimated); Study Completion 2020-07-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Retention in Treatment | Measured throughout 365 day duration of anticipated length of stay
  Participation in In-Home Addiction Treatment Program using length of stay reports
Brief Addiction Monitor questionnaire | Conducted monthly throughout 365 day anticipated length of stay in program
  Measure change in client report of symptoms related to substance use disorder
Positive Outcomes Measures Survey | Completed at week 3 or 4, Week 30, Week 35, Week 44, and Week 50 throughout 52 week anticipated length of program participation
  Measures changes in quality of life using client self-report inquiring about employment, connection to care team, community engagement using yes/no/not applicable response scale

SECONDARY OUTCOMES:
Relapse rates | Randomly administered throughout 365 day anticipated length of program participation
  Occurrence of substance use measured through urine drug screening and breathalyzer tests
Hospitalization | Measured throughout 365 day anticipated length of program participation
  Occurrence of Emergency Room and Inpatient hospital admissions
Detox and Residential Admissions | Measured throughout 365 day anticipated length of program participation
  Occurrence of residential treatment and detox admission

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kaiser, MS Ed, LPN, Principal Investigator — In-Home Addiction Treatment Institute, Inc.
Locations (1):
- Aware Recovery Care, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No